CLINICAL TRIAL: NCT01700257
Title: Different Strategies Using Autoantibodies and/or CT Scan Detection of Lung Cancer
Brief Title: Lung Cancer Screening Study With Low-dose CT Scan and Blood Biomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Oncimmune-2550
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: High Risk of Developing Lung Cancer
Keywords: Lung cancer screening; Smokers or former smokers; Family history of lung cancer
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT scan & Early CDT Lung test (Other): Every study participant receives a CT scan & Early CDT-Lung test (biomarker blood test) for lung cancer screening purposes.
  Interventions: Radiation: CT scan & Early CDT Lung test; Other: CT scan & Early CDT Lung test

INTERVENTIONS:
Radiation: CT scan & Early CDT Lung test
  Other Names: Every study participant receives a CT scan & Early CDT-Lung test (biomarker blood test); for lung cancer screening purposes
Other: CT scan & Early CDT Lung test
  Other Names: CT scan & Early CDT-Lung test (biomarker blood test)for lung cancer screening.

SUMMARY:
Lung cancer is the number one cancer killer in the USA. Early stage lung cancer is asymptomatic. Most patients with lung cancer are usually symptomatic at diagnosis and already have advanced stage disease. Low dose CT screening (LDCT) for high risk individuals has recently been shown to decrease lung cancer mortality by 20%. However, 4 out of 5 lung cancer deaths are not prevented with LDCT screening alone.

DETAILED DESCRIPTION:
In this trial, the addition of a blood biomarker test is being combined with early LDCT to determine if screening with combination may result in detection of more lung cancer at an earlier stage of disease.The study will also assess if the blood test is able to detect lung cancers in high risk individuals when the LDCT is negative for cancer. There will be health-economic costs included in the final analysis of study data.

ELIGIBILITY:
Inclusion Criteria:

* Smokers or former smokers
* At least 20 pack year history of smoking
* Ages 50 - 75

Exclusion Criteria:

* Had a CT scan of chest within last 24 months
* History of any cancer within 10 yrs (except skin cancer or cervical cancer)
* A serious illness that decreases life expectancy to less than 5 years
* Any current use of Oxygen
* Uncontrolled congestive heart failure or cardiac arrhythmia that would prevent surgery for a lung lesion
* Severe COPD or dyspnea that would prevent lung surgery or stereotactic body radiotherapy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1361 (Actual)
Dates: Start 2012-05; Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
CT alone vs. both Early CDT-Lung test and CT scan. | One year
  Assess the number of lung cancers detected with CT alone vs. with both Early CDT-Lung test and CT scan. Compare positive CT results with positive/negative Early CDT Lung test results and assess ability of the combination to detect earlier stage lung cancer.

SECONDARY OUTCOMES:
Value of Early CDT-lung test in detecting cancer | One year
  Assess the value of Early CDT-lung test in detecting lung cancer in individuals who are CT scan negative but positive for Early CDT-lung.

OTHER OUTCOMES:
Health Economics | One Year
  Comparison of the health economic costs of Early CDT-Lung test and CT scan when each is used individually or in combination.

CONTACTS AND LOCATIONS:
Overall Officials: James R Jett, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States